CLINICAL TRIAL: NCT01406899
Title: Computer-Assisted Cognitive Behavior Therapy for Veterans With Substance Use Disorder
Brief Title: Computer-Based Training in Cognitive Behavior Therapy (CBT4CBT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JC0008
Record Dates: First submitted 2011-07-27; First posted 2011-08-01 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2012-03

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (No Intervention): Standard treatment as usual (TAU) in the VA Connecticut Healthcare System substance abuse clinic consisting of individual and group therapy sessions and regular urine monitoring.
- Computer-based treatment (Experimental): Standard treatment as usual (TAU) plus coping skills computer program. In addition to the individual and group therapy sessions (TAU), individuals will work with a computerized program that teaches skills for stopping substance use and increasing coping skills twice weekly for 8 weeks.
  Interventions: Behavioral: Computer Based Treatment

INTERVENTIONS:
Behavioral: Computer Based Treatment — Standard treatment as usual (TAU) plus coping skills computer program. In addition to the individual and group therapy sessions (TAU), individuals will work with a computerized program that teaches skills for stopping substance use and increasing coping skills twice weekly for 8 weeks.
  Other Names: Cognitive Behavioral Therapy
  Arms: Computer-based treatment

SUMMARY:
In this behavioral trial 80 substance abusing individuals will be randomly assigned to either treatment as usual in the substance abuse clinic of the Newington, CT VA hospital OR treatment as usual plus 8 hours of access to the 'CBT for CBT' computer program over a period of 8 weeks. Primary outcomes will be retention in treatment and reduction in substance use (percent days abstinent, confirmed by urine toxicology screens). The patients' ability to demonstrate coping skills through a computerized role-play evaluation will be a secondary outcome. A six-month follow-up will assess durability and/or delayed emergence of effects.

DETAILED DESCRIPTION:
This pilot study aims to evaluate the feasibility and effectiveness of adding a computer based training program in Cognitive Behavior Therapy ("CBT4CBT") for the treatment of addictions in a VA substance abuse outpatient clinic. Key secondary aims are to assess the impact of adding CBT4CBT to standard care on treatment attendance, engagement, retention, and to investigate if certain process measures are associated with substance use outcomes. Approximately 80 patients enrolled in the Newington Outpatient Substance Abuse Treatment Program (SATP) will be randomly assigned to either (A) treatment as usual, or (B) treatment as usual plus exposure to the CBT4CBT program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Recent (within 3 months) substance use
* meet current DSM-IV (Diagnostic and Statistical Manual-IV) criteria for substance use disorder
* fluent in English or at least a 6th grade reading level
* can commit to at least 8 weeks of treatment and willing to be randomized to treatment

Exclusion Criteria:

* Unstable housing situation
* Likelihood of going to prison during the intervention portion of study
* Recent opiate or benzodiazepine prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reduction in substance use | 8 weeks
  percent days abstinent, confirmed by urine toxicology screens

SECONDARY OUTCOMES:
Retention in treatment | 6 months
  did patient continued to be enrolled in substance abuse treatment at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, Ph.D., Study Director — Yale University
Locations (1):
- Connecticut VA Healthcare System, Newington, Connecticut, United States

REFERENCES:
- [Derived] Lichenstein SD, Kohler R, Ye F, Potenza MN, Kiluk B, Yip SW. Distinct neural networks predict cocaine versus cannabis treatment outcomes. Mol Psychiatry. 2023 Aug;28(8):3365-3372. doi: 10.1038/s41380-023-02120-0. Epub 2023 Jun 12. PMID 37308679